CLINICAL TRIAL: NCT04655430
Title: Effect of Application Time of 38% Silver Diamine Fluoride Solution on Arresting Dental Caries in Preschool Children: a Randomized Double Blinded Controlled Trial
Brief Title: Effect of Application Time of 38% Silver Diamine Fluoride Solution on Arresting Dental Caries in Preschool Childre
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun-Hung Chu, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKU20201127
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Early Childhood Caries
Keywords: silver diamine fluoride; application time; preschool children; early childhood caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 3-second SDF application (Experimental): 3-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 3-second SDF application
- 5-second SDF application (Experimental): 5-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 5-second SDF application
- 10-second SDF application (Experimental): 10-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 10-second SDF application
- 15-second SDF application (Experimental): 15-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 15-second SDF application
- 30-second SDF application (Experimental): 30-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 30-second SDF application
- 45-second SDF application (Experimental): 45-second application time of silver diamine fluoride (38% SDF) in arresting tooth decay (dental caries) in the primary teeth of preschool children.
  Interventions: Other: 45-second SDF application
- 60-second SDF application (Experimental): 60-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 60-second SDF application
- 120-second SDF application (Experimental): 120-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 120-second SDF application
- 180-second application time (Experimental): 180-second application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.
  Interventions: Other: 180-second SDF application

INTERVENTIONS:
Other: 3-second SDF application — Dosage: 3-second 38% SDF solution application
  Arms: 3-second SDF application
Other: 5-second SDF application — Dosage: 5-second 38% SDF solution application
  Arms: 5-second SDF application
Other: 10-second SDF application — Dosage: 10-second 38% SDF solution application
  Arms: 10-second SDF application
Other: 15-second SDF application — Dosage: 15-second 38% SDF solution application
  Arms: 15-second SDF application
Other: 30-second SDF application — Dosage: 30-second 38% SDF solution application
  Arms: 30-second SDF application
Other: 45-second SDF application — Dosage: 45-second 38% SDF solution application
  Arms: 45-second SDF application
Other: 60-second SDF application — Dosage: 60-second 38% SDF solution application
  Arms: 60-second SDF application
Other: 120-second SDF application — Dosage: 120-second 38% SDF solution application
  Arms: 120-second SDF application
Other: 180-second SDF application — Dosage: 180-second 38% SDF solution application
  Arms: 180-second application time

SUMMARY:
To determine the optimal application time of silver diamine fluoride (38% SDF) in arresting dental caries in the primary teeth of preschool children.

DETAILED DESCRIPTION:
Methods: The randomized double blinded clinical trial will recruit 414 healthy kindergarten children aged 3-5 years old with caries and with parental consent. The sample size is sufficient for the appropriate statistical analyses. The children will receive 0.004 mL 38% SDF (typical amount applied per manufacturer's instructions) to treat each caries lesion. The children will be classified into high and low caries rates and equably allocated into nine groups of SDF application time: 3, 5, 15, 30, 45, 60, 120 and 180 seconds. The children will be followed up for 6-months in their kindergartens. Clinical examinations after 6-months will be conducted to assess whether the caries is arrested. Information on confounding factors, such as oral hygiene habits and the use of other fluoride agents, will be collected through a parental questionnaire at the baseline and 6-months follow-up. The examiner, the children and the children's parents will be blind to the treatment allocation. The analysis will determine the significance of differences between the means of arrested caries at the various follow-ups; and Cochran-Armitage test will be used to evaluate the exposure (SDF-application time) to response relationship.

Significance: This study will help determine the optimal application time in SDF treatment. The study provides an evidence-based protocol for the use of silver diamine fluoride to arrest tooth decay in primary teeth of young children.

ELIGIBILITY:
Inclusion Criteria:

(a) 3-5 year old children attending the first to the third year of kindergarten; (b) free from any systemic conditions and generally healthy; (c) parents sign informed consent (d) having at least 1 tooth with cavitated dentine carious lesion.

Exclusion Criteria:

* uncooperative and difficult to manage, have major systemic diseases such as porphyria, or are on long-term medication such as anti-epileptic drugs.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 600 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The visible plaque index (VPI). | at 6-months follow-up
  Two areas (buccal and lingual) of each of the six index teeth (55/51/63/71/75/83) will be examined and recorded (presence/absence) without visible plaque.
dmft index | at 6-months follow-up
  The tooth discoloration, tooth status (decayed, missing or filled teeth teeth (dmft) index) and tooth mobility

CONTACTS AND LOCATIONS:
Locations (1):
- Local kindergartens, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan IG, Zheng FM, Sun IG, Lo ECM, Duangthip D, Chu CH. A Randomized Controlled Trial of Silver Diamine Fluoride Application Time. J Dent Res. 2025 Dec;104(13):1453-1461. doi: 10.1177/00220345251345801. Epub 2025 Jun 29. PMID 40583169
- [Derived] Yan IG, Zheng FM, Gao SS, Duangthip D, Lo ECM, Chu CH. Effect of application time of 38% silver diamine fluoride solution on arresting early childhood caries in preschool children: a randomised double-blinded controlled trial protocol. Trials. 2022 Mar 15;23(1):215. doi: 10.1186/s13063-022-06130-1. PMID 35292085